CLINICAL TRIAL: NCT00004700
Title: Phase II Long Term, Randomized Study of Recombinant Human Insulin-like Growth Factor I in Children With Hyperinsulinism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13382; CHP-FDR001181-DBPC
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-03

CONDITIONS: Hyperinsulinism
Keywords: endocrine disorders; hyperinsulinism; rare disease
MeSH Terms: conditions — Hyperinsulinism; Endocrine System Diseases; Rare Diseases | interventions — Insulin-Like Growth Factor I

INTERVENTIONS:
Drug: insulin-like growth factor I

SUMMARY:
OBJECTIVES:

Evaluate the safety and efficacy of long term recombinant human insulin-like growth factor I in children with hyperinsulinism.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, cross-over study.

Patients are randomized to receive recombinant human insulin-like growth factor I (IGF-I) or placebo subcutaneously twice daily for 4 weeks. After a 2 week washout period, patients are crossed over to the other regimen for an additional 4 weeks.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Diagnosis of hyperinsulinism (i.e., evidence of fasting hypoglycemia with inadequate suppression of insulin, normal pituitary and adrenal function, and increased insulin action) Suboptimal control of blood sugar (i.e., inability to fast at least 10 hours with a blood sugar of 60 mg/dL or greater) --Prior/Concurrent Therapy-- See Disease Characteristics --Patient Characteristics-- Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other major medical conditions No known adverse reaction to recombinant human insulin-like growth factor I

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16
Dates: Start 1995-08; Study Completion 1999-01

CONTACTS AND LOCATIONS:
Overall Officials: Pinchas Cohen, Study Chair — Children's Hospital of Philadelphia